CLINICAL TRIAL: NCT03638778
Title: A Trial Comparing Exposure of Semaglutide When Dosing New Formulations of Oral Semaglutide to Healthy Male Subjects
Brief Title: Research Study Comparing Different Tablets With the Study Medicine Semaglutide in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4427; U1111-1206-6210 (Other: World Health Organization (WHO)); 2017-005023-24 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2018-08-08; First posted 2018-08-20 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Oral semaglutide (reference) (Active Comparator): Participants will receive oral semaglutide (reference) for 10 days.
  Interventions: Drug: Semaglutide 3 mg; Drug: Semaglutide 7 mg
- Oral semaglutide formulation B (Experimental): Participants will receive oral semaglutide formulation B for 10 days.
  Interventions: Drug: Semaglutide B 3 mg; Drug: Semaglutide B 7 mg
- Oral semaglutide formulation C (Experimental): Participants will receive oral semaglutide formulation C for 10 days.
  Interventions: Drug: Semaglutide C 3 mg; Drug: Semaglutide C 7 mg
- Oral semaglutide formulation D (Experimental): Participants will receive oral semaglutide formulation D for 10 days.
  Interventions: Drug: Semaglutide D 3 mg; Drug: Semaglutide D 7 mg

INTERVENTIONS:
Drug: Semaglutide 3 mg — Semaglutide 3 mg will be administered once daily (OD) orally in the morning from day 1 to 5.
  Arms: Oral semaglutide (reference)
Drug: Semaglutide 7 mg — Semaglutide 7 mg will be administered OD orally in the morning from day 6 to 10.
  Arms: Oral semaglutide (reference)
Drug: Semaglutide B 3 mg — Semaglutide B 3 mg will be administered OD orally in the morning from day 1 to 5.
  Arms: Oral semaglutide formulation B
Drug: Semaglutide B 7 mg — Semaglutide B 7 mg will be administered OD orally in the morning from day 6 to 10.
  Arms: Oral semaglutide formulation B
Drug: Semaglutide C 3 mg — Semaglutide C 3 mg will be administered OD orally in the morning from day 1 to 5.
  Arms: Oral semaglutide formulation C
Drug: Semaglutide C 7 mg — Semaglutide C 7 mg will be administered OD orally in the morning from day 6 to 10.
  Arms: Oral semaglutide formulation C
Drug: Semaglutide D 3 mg — Semaglutide D 3 mg will be administered OD orally in the morning from day 1 to 5.
  Arms: Oral semaglutide formulation D
Drug: Semaglutide D 7 mg — Semaglutide D 7 mg will be administered OD orally in the morning from day 6 to 10.
  Arms: Oral semaglutide formulation D

SUMMARY:
This study looks at different tablets with a new study medicine called semaglutide. It is to treat diabetes. The aim of the study is to find out how much study medicine from 4 different tablets is taken up in the body. Participants will either get semaglutide in the tablet currently being studied in large studies, or 1 of the 3 new tablets that also contains 'semaglutide' - which treatment participants get is decided by chance. The tablet version of study medicine is a new medicine that cannot be prescribed. Semaglutide can be prescribed as injections for the treatment of diabetes in some countries. Participants will get 1 tablet per day for 10 days. The tablets should be taken in the morning by mouth together with half a glass of water. After dosing participants have to wait 30 minutes before participants may eat or drink. The study will last up to 70 days. Participants will have 17 clinic visits with the study doctor. Some of the visits are overnight stays. Participants will have blood tests at every visit.

ELIGIBILITY:
Inclusion Criteria: - Male, aged 18-64 years (both inclusive) at the time of signing informed consent. - Body mass index (BMI) between 20.0 and 29.9 kg/m^2 (both inclusive). - Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator. Exclusion Criteria: - Glycated haemoglobin (HbA1c) greater than or equal to 6.5% (48 mmol/mol) at screening. - Use of tobacco and nicotine products, defined as any of the below: a) Smoking more than 5 cigarettes or the equivalent per day. b) Not willing to refrain from smoking and use of nicotine substitute products during the in-house period(s). - History* of major surgical procedures involving the stomach potentially affecting absorption of trial products (e.g., subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery). - Presence of clinically significant gastrointestinal disorders or symptoms of gastrointestinal disorders potentially affecting absorption of drugs or nutrients, as judged by the investigator. - Personal or first degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma*. - History* or presence of pancreatitis (acute or chronic). *As declared by subject.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
AUC0-24h,sema,day10, area under the semaglutide plasma concentration time curve from 0 to 24 hours after the 10th dosing | 0 to 24 hours on day 10
  Calculated based on semaglutide measured in blood.

SECONDARY OUTCOMES:
Cmax,sema,day10, maximum observed semaglutide plasma concentration from 0 to 24 hours after the 10th dosing | 0 to 24 hours on day 10
  Calculated based on semaglutide measured in blood.
tmax,sema,day10, time to maximum observed semaglutide plasma concentration from 0 to 24 hours after the 10th dosing | 0 to 24 hours on day 10
  Calculated based on semaglutide measured in blood.
AUC0-30min,sema,day10, area under the semaglutide plasma concentration time curve from 0 to 30 minutes after the 10th dosing | 0 to 30 minutes on day 10
  Calculated based on semaglutide measured in blood.
t½,sema,day10, terminal half-life of semaglutide up to 35 days after the 10th dosing | Days 10-45
  Calculated based on semaglutide measured in blood. Measured from the 10th. dosing (on Day 10) and up to 35 days after the 10th. dosing (i.e. Day 45).
Number of treatment emergent adverse events | Days 1-47
  Count of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com/sharing-results